CLINICAL TRIAL: NCT04588714
Title: Feasibility and Preliminary Effects of the Resilience-based, Energy Management to Enhance Wellbeing in Systemic Sclerosis (RENEW) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Susan Murphy, Associate Professor of Physical Medicine and Rehabilitation and Research Associate Professor, Institute of Gerontology, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00186877
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Scleroderma
Keywords: Peer mentor; Web-based
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: Pilot study, one arm, pre-test, post-test trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resilience-based, Energy Management to Enhance Wellbeing (RENEW) (Experimental): RENEW is a 12-week program in which participants are paired with a peer mentor who serves as their health coach throughout the intervention period. The website serves as the program "workbook" to help promote skill practice and attainment in areas like goal setting, pacing, relaxation, etc.
  Interventions: Behavioral: Resilience-based, Energy Management to Enhance Wellbeing (RENEW)

INTERVENTIONS:
Behavioral: Resilience-based, Energy Management to Enhance Wellbeing (RENEW) — The program includes unlimited website access and 10 scheduled phone calls with an assigned peer mentor.

SUMMARY:
Researchers are testing a web-based peer-led program to help manage energy and symptoms in people who have scleroderma. Resilience-based, Energy Management to Enhance Wellbeing (RENEW) was created by researchers, doctors, and patients with scleroderma. The goal is to help people with scleroderma feel better.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of systemic sclerosis including:

  * Diffuse or limited cutaneous
* Have access to a reliable, internet-connected device (e.g. computer, tablet)
* Be able to read, speak, and understand English
* Participants need to report a score of at least 4 on a scale of 0 - 10 of fatigue severity, a cut-off for at least moderate fatigue in other fatiguing conditions.

Exclusion Criteria:

* Complex, unstable health issues that would preclude full participation in the study
* Planning to start new treatment for fatigue, pain, mood during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by intervention participant retention | 12 weeks
  Number of participants who complete the study
Feasibility as assessed by the participation in intervention related phone calls | 12 weeks
  Number of completed peer-mentor calls

SECONDARY OUTCOMES:
Feasibility as assessed by active participant involvement | 12 weeks
  Number of minutes spent accessing the RENEW website/app
Feasibility as assessed by the peer mentor health coach time | 12 weeks
Feasibility as assessed by the time spent in preparation for intervention phone calls | 12 weeks
  Preparation time of peer mentors will be documented in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Murphy, ScD, OTR/L, Principal Investigator — University of Michigan; Dinesh Khanna, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No